ImmunityBio, Inc.

# THEMBA II T-CELL VACCINE: A PHASE 1/2 STUDY OF THE SAFETY, REACTOGENICITY, AND IMMUNOGENICITY OF VACCINATION WITH saRNA COVID-19 VACCINES

| Study Number: | COVID-4.015 |
|---|---|
| IND Sponsor: | ImmunityBio, Inc. |
| National Principal Investigator | Professor Shabir A. Madhi South African Medical Research Council Vaccines and Infectious Diseases Analytics Research Unit Wits Health Consortium (A subsidiary of the University of the Witwatersrand) Johannesburg, South Africa shabir.madhi@wits ac za |
| Sponsor Contact: (For medical questions/emergencies) | Lennie Send r MD Medical Monitor 9920 Jefferson Blvd Culver City CA 90232 Email: lennie.sender@immunitybio.com Cell Phone: 714-615-2350 |

| Protocol Version | Date |
|------------------|------------------|
| Version 1 | 21 January 2022 |
| Version 2 | 17 February 2022 |
| Version 3 | 17 March 2022 |
| Version 4 | 27 October 2022 |

ImmunityBio, Inc.

Clinical Trial Protocol: COVID-4.015 Version 4

#### STATEMENT OF COMPLIANCE

This trial will be conducted in accordance with applicable local regulatory requirements, Good Clinical Practice (GCP) as described in the International Conference on Harmonization (ICH) Guideline for GCP (E6 [R2]), United States (US) Code of Federal Regulations (CFR) applicable to clinical studies and the general ethical principles outlined in the Declaration of Helsinki. The study will receive approval from an Institutional Review Board (IRB) or Independent Ethics Committee (IEC) prior to commencement. The Principal Investigator will assure that no deviation from, or changes to the protocol will take place without prior agreement from the sponsor and documented approval from the IRB/IEC, except where necessary to eliminate an immediate hazard(s) to the trial participants.

I agree to ensure that all staff members involved in the conduct of this study are informed about their obligations in meeting the above commitments.

| Signed: | Date: |
|---------|-------|

ImmunityBio, Inc.


#### PROTOCOL SYNOPSIS

#### Name of Sponsor/Company:

ImmunityBio, Inc.

#### Name of Investigational Products:

- 1. AAHI -SC2 self-amplifying RNA (saRNA) against SARS-CoV-2 Spike protein delivered by nanostructured lipid carrier (NLC) Vaccine
- 2. AAHI-SC3 self-amplifying RNA (saRNA) against SARS-CoV-2 nucleocapsid protein delivered by nanostructured lipid carrier (NLC) Vaccine

Note that AAHI-SC3 is now comprised of saRNA against SARS-CoV-2 nucleocapsid protein only while in previous versions of this protocol, AAHI-SC3 was comprised of saRNA against SARS-CoV-2 nucleocapsid and Spike proteins.

#### Name of Active Ingredients:

- 1. AAHI-SC2 Vaccine
- 2. AAHI-SC3 Vaccine

#### **Title of Study:**

Themba II T-Cell Vaccine: A phase 1/2 Study of the Safety, Reactogenicity, and Immunogenicity of Vaccination with saRNA COVID-19 Vaccines

#### **Study Number:**

COVID-4.015

## **Study Phase:**

Phase 1/2

| C4 1 | $\alpha$ | |
|-------|----------|---------|
| Study | On | ectives |

**Study Endpoints** 

#### Phase 1

#### **Phase 1 Primary Objective**

<u>Safety</u>: To determine the safety and reactogenicity of homologous and heterologous vaccination with saRNA COVID-19 vaccines.

- Incidence of medically-attended adverse events (MAAEs) and serious adverse events (SAEs) through 1 week post final vaccine administration
- Incidence of MAAEs and SAEs through 30 days post final vaccine administration
- Incidence of MAAEs and SAEs through
   6 months post final vaccine administration
- Incidence and severity of solicited local reactogenicity AEs through 1 week after each vaccine dose
- Incidence and severity of solicited systemic reactogenicity AEs through 1 week after each vaccine dose

ImmunityBio, Inc.

 Incidence and severity of unsolicited AEs through 1 week post final vaccine administration

Incidence and severity of unsolicited AEs through 30 days post final vaccine administration
Incidence of abnormal changes of laboratory safety examinations

Changes in vital signs

#### **Phase 1 Secondary Objective**

Immunogenicity: To determine immunogenicity of homologous and heterologous vaccination with saRNA COVID-19 vaccines, as determined by changes in humoral and cellular response.

Humoral Immunogenicity:

- Geometric mean titer (GMT) of S-specific and N-specific IgG antibodies against 2019 novel coronavirus tested by ELISA in serum
- GMT of neutralizing antibody

Cellular Immunogenicity:

 T cell activity against SARS-CoV-2 S protein and N protein as assayed by ELISpot

#### Phase 2

#### **Phase 2 Primary Objective**

Immunogenicity: To determine immunogenici y of homologous and heterologous vaccination with saRNA COVID-19 vaccines, as determin d by changes in humoral and cellular response

Humoral Immunogenicity:

- GMT of S-specific and N-specific IgG antibodies against 2019 novel coronavirus tested by ELISA in serum
- GMT of neutralizing antibody

Cellular Immunogenicity:

 T cell activity against SARS-CoV-2 S protein and N protein as assayed by the ELISpot assay

#### **Phase 2 Secondary Objectives**

<u>Safety:</u> To determine the safety and reactogenicity of homologous and heterologous vaccination with saRNA COVID-19 vaccines.

- Incidence of MAAEs and SAEs through 30 days post final vaccine administration
- Incidence of MAAEs and SAEs through 6 months post final vaccine administration
- Incidence and severity of solicited local reactogenicity AEs through 1 week after each vaccine dose
- Incidence and severity of solicited systemic reactogenicity AEs through 1 week after each vaccine dose






ImmunityBio, Inc.

#### **Study Design:**

This is a phase 1/2 open-label study assessing the safety, reactogenicity, and immunogenicity of saRNA COVID-19 boost vaccines in participants that have been previously vaccinated against or previously infected with COVID-19. Participants enrolled will include individuals previously vaccinated against COVID-19 or previously infected with COVID-19 > 3 months prior to enrollment. Previously unvaccinated/vaccinated status and previously uninfected/infected status will be established by medical history and by SARS-CoV-2 serology assessed in the prescreening visit.

The phase 1 study is a single arm, open-label study. The phase 2 and study is a randomized open-label study. For the phase 2 study, laboratory analyses of immunogenicity assessments will be performed blind to participants' vaccine treatment on study. In all study phases, SARS-CoV-2 serological status will be assessed in a prescreening visit.

Participants will be  $\geq 18$  years of age who are healthy or have medically-stable chronic diseases. The treatment regime is described in the sections that follow. The study schema is shown in Figure 1.

#### Phase 1

In the phase 1 study, up to 60 previously vaccinated/infected participants will be enrolled in 6 separate cohorts to receive a single vaccine boost consisting of either the AAHI-SC2 or AAHI-SC3 vaccines. Dosing schedule, mode of administration, and dosage for phase 1 are indicated in the table below.

| Phase | Cohort | Participants | Vaccine | D sing<br>Schedule | Dosage |
|-------|--------|--------------|----------|--------------------|----------|
| SE 1 | 1A | 10 | AAHI-SC2 | Day 1 | 25 μg IM |
| | 1B | 10 | AAHI-SC2 | Day 1 | 50 μg IM |
| | 1C | 10 | AAHI-SC2 | Day 1 | 70 μg IM |
| PHASE | 2A | 10 | AAHI-SC3 | Day 1 | 25 μg IM |
| | 2B | 10 | AAHI-SC3 | Day 1 | 50 μg IM |
| | 2C | 10 | AAHI-SC3 | Day 1 | 85 μg IM |

Safety will be assessed for all participants and will include monitoring of vital signs, and incidence and severity of AEs. Blood samples will be collected for hematology and chemistry analyses and urine samples will be collected for urinalysis. Toxicities will be graded using the Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (2007).

For each cohort in phase 1, after all 10 participants have completed the toxicity assessment period, the SRC will review safety results to determine if the event warrants stopping the trial, modifying the trial, or continuing without modification.

Solicited local and systemic reactogenicity AEs will be collected using diaries for 7 days following study intervention (ie, administration of vaccine). Unsolicited AEs will be recorded in a diary from time of vaccination until 30 days after study intervention. MAAEs and SAEs will be recorded for 6 months after study intervention (related MAAEs and SAEs will be recorded at any time).

Immunogenicity analyses will be conducted by collecting serum and peripheral blood mononuclear cell (PBMC) samples from individual participants before and after vaccinations to test for humoral- and cell-mediated immune responses. Neutralizing antibodies will be assessed.


ImmunityBio, Inc.

#### Phase 2

In the phase 2 study, up to 120 previously vaccinated/infected additional participants will be enrolled. Participants in phase 2 will be randomized 1:1:1:1 to receive Janssen or Pfizer-BioNTech vaccine (control arm), the AAHI-SC2 vaccine (experimental arm 1), or the AAHI-SC3 vaccine (experimental arms 2 and 3). Dose levels for the AAHI-SC2 and AAHI-SC3 vaccines will be as determined in the phase 1 study. Randomization will be stratified by age (18 to 55 years or > 55 years), by previous infection (previously infected or not), and by HIV status (positive or negative). Treatment arms are shown in the table below:

| Treatment Arm | Participants | Vaccine | Dosing schedule | Dosage |
|---|---|---|---|---|
| Control arm | 30 | Emergency Use Authorization (EUA) or approved vaccine | | Per prescribing information |
| Experimental arm 1 | 30 | AAHI-SC2 | Day 1 | TBD: As determined in phase 1 study |
| Experimental arm 2 | 30 | AAHI-SC3 | Day 1 | TBD: As determined in phase 1 study |
| Experimental arm 3 | 30 | AAHI-SC3 | Day 1 and<br>day 29 | TBD: As determined in phase 1 study |

In addition to dosing visits described above, all participants in all phases of the study will have follow-up study visits for data collection.

The SRC will provide ongoing safety review in the phase 2 study. If a possible safety signal is detected, the SRC will determine if the event warrants stopping the trial, modifying the trial, or continuing without modification.

Solicited local and systemic reactogenicity AEs will be collected using diaries for 7 days following study intervention (ie, administration of vaccine). Unsolicited AEs will be recorded in a diary from time of vaccination until 30 days after study intervention. MAAEs and SAEs will be recorded for 6 months after study intervention (related MAAEs and SAEs will be recorded at any time).

Immunogenicity analyses will be conducted by collecting serum and PBMC samples from individual participants before and after vaccinations to test for humoral- and cell-mediated immune responses. Neutralizing antibodies will be assessed.

#### **Enrollment (planned):**

Initially up to 180 participants will be enrolled in this study (60 participants in phase 1 and 120 participants in phase 2).

#### **Eligibility Criteria:**

#### **Inclusion Criteria:**

- 1. Healthy adults  $\geq$  18 years of age at time of enrollment.
- 2. Vaccinated with an EUA or approved vaccine against COVID-19  $\geq$  3 months prior to enrollment on study or infection with COVID-19  $\geq$  3 months prior to enrollment on study.
- 3. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.


ImmunityBio, Inc.

- 4. Agrees to the collection of biospecimens (eg, nasopharyngeal [NP] swabs) and venous blood per protocol.
- 5. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
- 6. Temperature < 38°C.
- 7. Agreement to practice effective contraception for female participants of childbearing potential and non-sterile males. Female participants of childbearing potential must agree to use effective contraception while on study until at least 1 month after the last dose of vaccine. Non-sterile male participants must agree to use a condom while on study until at least 1 month after the last dose of vaccine. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm), intrauterine devices (IUDs), oral contraceptives, injectable contraceptives, patches, implants and abstinence.
- 8. HIV-positive participants must have been on anti-retroviral therapy for  $\geq 4$  weeks and have HIV-1 viral load < 1,000 copies/mL at the time of enrollment.

#### **Exclusion Criteria:**

- 1. Serious adverse reaction to any vaccine, any unrelated medication or any component of the investigational vaccine, including a history of anaphylaxis and symptoms of a severe allergic reaction and history of allergies in the past.
- 2. Confirmed current COVID-19, previous SARS-CoV-2 infection in the last < 3 months, or PCR positive for SARS-CoV-2 at screening
- 3. Vaccinated with an EAU-approved vaccine against COVID-19 in the last < 3 months.
- 4. Pregnant or breastfeeding women
- 5. Any participants with a history of myocarditis or pericarditis.
- 6. Chronic lung disease (included COPD) as evidenced by one or more exacerbations requiring a course of steroids in the last year, or the requiring chronic low dose oral steroids to prevent exacerbations. Uncontrolled asthma, defined as requiring reliever inhaler (short-acting beta agonist or ipratropium bromide) more than twice a week is also excluded.
- 7. Bone marrow or organ transplant recipient
- 8. Extreme obesity (defined as BMI of 40 kg/m<sup>2</sup> or higher).
- 9. Chronic kidney disease requiring dialysis.
- 10. History of liver disease.
- 11. Any disease associated with acute fever, or any infection.
- 12. Participants with acquired or hereditary immunodeficiencies other than well-controlled HIV are excluded from enrollment.
- 13. Current diagnosis of active tuberculosis.
- 14. History of hereditary, idiopathic or acquired angioedema.


ImmunityBio, Inc.

- 15. No spleen or functional asplenia.
- 16. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon (IFN), or immunomodulators. The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
- 17. According to the judgement of the investigator any medical, psychiatric, psychological, social, occupational or other conditions that could affect the participants ability to sign informed consent, provide safety assessment data or comply with the requirements of the study protocol.
- 18. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

#### **Duration of Treatment:**

For most participants, treatment will be confined to study day 1. For participants in experimental arm 3 of the phase 2 study, treatment will occur on day 1 and day 29.

#### **Duration of Follow-up:**

Participants who receive study treatment will be followed by a health care professional until either death (by any cause) or for 1 year past first administration of vaccine.

#### Reference Therapy, Dosage, and Mode of Administration:

Janssen or Pfizer-BioNTech vaccine.

#### **Evaluation of Endpoints:**

**Safety:** Safety endpoints include assessments of treatment-emergent MAAEs, SAEs, reactogenicity AEs, unsolicited AEs, safety laboratory tests and vital signs. Toxicities will be graded using the Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (2007).

**Immunogenicity:** Immunogenici y endpoints will include GMT of IgG binding antibodies and GMT of neutralizing antibodies. T-Cell activity against SARS-CoV-2 will be assessed.

#### **Statistical Methods:**

The purpose of this phase 1/2 study is to determine the safety, reactogenicity, and immunogenicity of saRNA COVID-19 boost vaccines in participants that have been previously vaccinated against or previously infected with COVID-19. Participants enrolled will include individuals previously vaccinated against COVID-19 or previously infected with COVID-19 > 3 months prior to enrollment.

The phase 1 study is a single arm, open-label study. The phase 2 study is a randomized open-label study. For the phase 2 study, laboratory analyses of immunogenicity assessments will be performed blind to participants' vaccine treatment on study. Results for phase 1 will be summarized by cohort and results for phase 2 will be summarized for each randomized arm.

Descriptive statistics will be presented for all study endpoints. No statistical comparisons of the phase 2 arms is planned.

**Safety Analyses:** Safety will be assessed by the incidence of treatment-emergent MAAEs, SAEs, and solicited local and systemic reactogenicity AEs, and unsolicited AEs for the time period of interest, overall and by grade using the Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (2007). Clinically significant changes in safety laboratory tests and vital signs also will be summarized.

ImmunityBio, Inc.


**Immunogenicity Analyses:** GMTs and their associated 95% confidence intervals (CIs) will be computed by exponentiation of the corresponding log-transformed means and 95% CIs. T cell activity will be summarized.



Figure 1: Study Schema – Previously Vaccinated/Infected Participants



## Clinical Trial Protocol: COVID-4.015 Version 4

## **TABLE OF CONTENTS**

| TITLE PA | AGE | |
|---|---|---|
| STATEM | IENT OF COMPLIANCE | |
| PROTOC | COL SYNOPSIS | |
| LIST OF | ABBREVIATIONS AND DEFINITIONS OF TERMS | 19 |
| 1. | BACKGROUND AND STUDY RATIONALE | 22 |
| 1.1. | SARS-CoV-2 and COVID-19 | 22 |
| 1.2. | Study Rationale | 22 |
| 1.2.1. | Rationale for Self-Amplifying RNA Vaccine Vectors | 2 |
| 1.2.2. | Rationale for Revised Version of AAHI-SC3 Product | 22 |
| 1.3. | AAHI-SC2 Vaccine | 2 |
| 1.3.1. | Physical, Chemical, and Pharmaceutical Properties and Formulations | 2 |
| 1.3.1.1. | saRNA | 2 |
| 1.3.1.2. | Nanostructured Lipid Carrier (NLC) Formulation | 2 |
| 1.3.1.3. | Storage and Administration | |
| 1.3.2. | Nonclinical Experience | 24 |
| 1.3.2.1. | In Vivo Safety and Immunogenicity of AAHI-SC2 in Mice | 2 |
| 1.3.2.2. | In Vivo Immunogenicity of Homologous or Heterologous Vaccination With AAHI-SC2 Prime and hAd5-S-Fusion+N-ETSD Boost in Mice | 2 |
| 1.3.2.3. | In Vivo Safety, Immunog nicity, and Protection Studies of saRNA/NLC in Nonhuman Primates | 3 |
| 1.3.2.4. | In Vivo Safety and Immunogenicity of saRNA/NLC Targeted Against Cancer Neoantigens in Nonhuman Primates | 32 |
| 1.3.2.5. | In Vivo Repeat Dose Toxicity and Biodistribution Study of AAHI-SC2 in New Zealand White Rabbits | 3 |
| 1.3.2.6. | In Vivo Immunogenicity and Protective Efficacy of AAHI-SC2 in Nonhuman Primates | 3′ |
| 1.3.3. | Clinical Experience | 3 |
| 1.4. | AAHI-SC3 Vaccine | 3 |
| 1.4.1. | Physical, Chemical, and Pharmaceutical Properties and Formulations | 3 |
| 1.4.1.1. | saRNA | 3 |
| 1.4.1.2. | Nanostructured Lipid Carrier (NLC) | 39 |
| 1.4.1.3. | Storage and Administration | 39 |
| 1.4.2. | Nonclinical Experience with AAHI-SC3 Vaccine | 39 |

## ImmunityBio, Inc.

| 1.4.2.1. | In Vivo Immunogenicity Studies in Mice | 39 |
|----------|----------------------------------------|----|
| 1.4.3. | Clinical Experience | |
| 1.5. | Rationale for Starting Doses | |
| 1.6. | Potential Risks and Benefits | |
| 1.6.1. | Potential Risks | 43 |
| 1.6.1.1. | saRNA and NLC Vaccine Platform | 43 |
| 1.6.1.2. | AAHI-SC2 Vaccine | 43 |
| 1.6.1.3. | AAHI-SC3 Vaccine | 43 |
| 1.6.2. | Potential Benefits | 43 |
| 1.6.2.1. | saRNA and NLC Vaccine Platform | |
| 1.6.2.2. | AAHI-SC2 Vaccine | 43 |
| 1.6.2.3. | AAHI-SC3 Vaccine | 44 |
| 2. | STUDY OBJECTIVES | 45 |
| 2.1. | Phase 1 | |
| 2.1.1. | Primary Objective | 45 |
| 2.1.2. | Secondary Objective | 45 |
| 2.2. | Phase 2 | 45 |
| 2.2.1. | Primary Objective | |
| 2.2.2. | Secondary Objectives | 45 |
| 3. | INVESTIGATIONAL PLAN | 46 |
| 3.1. | Study Design | 46 |
| 3.2. | Number of Participants | 48 |
| 3.3. | Duration of Study | 48 |
| 3.3.1. | Duration of Treatment | 48 |
| 3.3.2. | Duration of Follow-Up | 48 |
| 3.3.3. | End of Study | 48 |
| 3.4. | Study Endpoints | 48 |
| 3.4.1. | Phase 1 | 48 |
| 3.4.1.1. | Primary Endpoints | 48 |
| 3.4.1.2. | Secondary Endpoints | 49 |
| 3.4.2. | Phase 2 | |
| 3.4.2.1. | Primary Endpoints | 49 |

## ImmunityBio, Inc.

| 3.4.2.2. | Secondary Endpoints | 49 |
|---|---|---|
| 4. | PARTICIPANT ENROLLMENT AND WITHDRAWAL | 50 |
| 4.1. | Participant Eligibility | 50 |
| 4.1.1. | Inclusion Criteria | 50 |
| 4.1.2. | Exclusion Criteria | 50 |
| 4.2. | Strategies for Recruitment and Retention | 51 |
| 4.3. | Screen Failures | 51 |
| 4.4. | Withdrawal of Participants | 52 |
| 4.5. | Treatment Discontinuation | 52 |
| 4.6. | Replacement of Participants | |
| 4.7. | Premature Termination or Suspension of Study | 52 |
| 5. | TREATMENT PROCEDURES | 53 |
| 5.1. | Investigational Product Dosage, Route of Administration, and Dosing Schedule | 53 |
| 5.1.1. | Formulation, Appearance, and Packaging | |
| 5.1.2. | Storage and Stability | 53 |
| 5.1.3. | Acquisition | 54 |
| 5.1.4. | Dose Preparation | 54 |
| 5.1.5. | Dosing and Administration | 54 |
| 5.1.6. | Accountability of IP | |
| 5.1.7. | Management of Adverse Events and Individual Stopping Criteria | 55 |
| 6. | STUDY PROCEDURES AND EVALUATIONS | 56 |
| 6.1. | Prescreening Assessments | 56 |
| 6.2. | Baseline/Screening Assessments | 56 |
| 6.3. | Safety Assessments | 57 |
| 6.3.1. | Solicited Local and Systemic Adverse Events | 57 |
| 6.3.2. | Unsolicited Adverse Events | 57 |
| 6.4. | Follow-Up for Disease History | 57 |
| 6.5. | Clinical Laboratory Procedures and Evaluations | 58 |
| 6.6. | Laboratory Procedures and Evaluations for Immunological Endpoints and Other Laboratory Procedures and Evaluations | 58 |
| 6.6.1. | Immunogenicity Assessments | 59 |
| 6.6.1.1. | Cellular and Humoral Response to SARS-CoV-2 Proteins | 59 |

## ImmunityBio, Inc.

| 6.6.2. | SARS-CoV-2 Testing | 59 |
|---|---|---|
| 6.6.3. | HIV Testing | 59 |
| 6.7. | Study Schedule | 59 |
| 6.7.1. | Screening Procedures and Evaluations | 59 |
| 6.7.1.1. | Medical History | 59 |
| 6.7.2. | Study Period(s) | 63 |
| 6.7.3. | End-of-Study Procedures and Evaluations | 63 |
| 6.8. | Concomitant Medications | 63 |
| 6.9. | Participant Access to Study Medications at Close of Study | 63 |
| 7. | ADVERSE EVENT MONITORING AND REPORTING | 64 |
| 7.1. | Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (2007) | 64 |
| 7.2. | Definition of Adverse Events | 70 |
| 7.3. | Definition of Serious Adverse Events | 71 |
| 7.4. | Evaluation of Adverse Events | |
| 7.4.1. | Severity/Intensity | 71 |
| 7.4.2. | Relationship to the Investigational Product | 72 |
| 7.4.3. | Duration of Adverse Events | 72 |
| 7.4.4. | Outcome | 73 |
| 7.5. | Reporting Procedures | |
| 7.5.1. | Reporting Procedures for Adverse Events | 73 |
| 7.5.2. | Reporting Procedures for Serious Adverse Events | 73 |
| 7.5.3. | Expedited Reporting of Adverse Events | 74 |
| 7.6. | Reporting of Pregnancy | 74 |
| 7.6.1. | Females of Childbearing Potential | 74 |
| 7.6.2. | Male Participants | 75 |
| 7.7. | Safety Queries | 75 |
| 7.8. | Safety Oversight | 75 |
| 7.8.1. | Safety Review Committee | 76 |
| 7.8.1.1. | Safety Review Committee Members | 76 |
| 7.8.2. | Phase 1 Study Toxicity Study Stopping Rules | 76 |
| 7.8.2.1. | Planned Safety Review Committee Meetings | 77 |

## ImmunityBio, Inc.

| 7.8.3. | Phase 2 Safety Review Committee Review | 77 |
|---|---|---|
| 8. | STATISTICAL CONSIDERATIONS | 78 |
| 8.4. | Sample Size | 79 |
| 9. | INVESTIGATOR RESPONSIBILITIES | 80 |
| 10. | REGULATORY CONSIDERATIONS | 81 |
| 10.1. | Good Clinical Practice | 81 |
| 10.2. | Participant Information and Informed Consent | 81 |
| 10.3. | Confidentiality | 81 |
| 10.4. | Protocol Amendment | 82 |
| 10.5. | Institutional Review Board/Independent Ethic Committee Review and Approval | 82 |
| 10.6. | Approval | 82 |
| 11. | DATA HANDLING AND RECORDKEEPING | |
| 11.1. | Data/Documents | 83 |
| 11.2. | Data Management | 83 |
| 11.3. | Inspection of Records | 83 |
| 11.4. | Retention of Records | 83 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | |
| 12.1. | Audits and Inspections | 85 |
| 13. | PUBLICATION POLICY | 86 |
| 14. | REFERENCES | 87 |
| APPENDIX | X 1. SAMPLE DIARY FOR SOLICITED EVENTS | 88 |
| APPENDIX | X 2. SAMPLE DIARY FOR UNSOLICITED EVENTS | 91 |
| APPENDIX | X 3. SPONSOR SIGNATURE | 92 |

ImmunityBio, Inc.

## **LIST OF TABLES**

| Γable 1: | Mouse Immunogenicity Study Treatment Groups | 25 |
|---|---|---|
| Гable 2: | Treatment Groups for Rabbit Toxicity and Biodistribution Study | 34 |
| Γable 3: | Mouse Immunogenicity Treatment Groups for Spike + Nucleocapsid Proteins | 39 |
| Гable 4: | Phase 1 Previously Vaccinated/Infected Dosing Schedule | 46 |
| Гable 5: | Phase 2 Previously Vaccinated/Infected Dosing Schedule | 47 |
| Гable 6: | Formulation, Appearance, and Packaging of Investigational Products | 53 |
| Гable 7: | Storage and Stability of Investigational Products | 53 |
| Гable 8: | Preparation of Investigational Product | 54 |
| Гable 9: | Laboratory Assessments | 58 |
| Гable 10: | Schedule of Events: Previously Vaccinated/Infect d Participants | 60 |
| Гable 11: | Clinical Abnormalities: Local Reaction to Injectable Products | 64 |
| Гable 12: | Clinical Abnormalities: Vital Signs | 65 |
| Гable 13: | Clinical Abnormalities: Systemic | 66 |
| Гable 14: | Laboratory Abnormalities: Serum | 67 |
| Гable 15: | Laboratory Abnormalities: Hematology | 69 |
| Table 16: | Laboratory Abnormalities: Urine | 70 |

## **LIST OF FIGURES**

| Figure 1: | Study Schema – Previously Vaccinated/Infected Participants | 11 |
|---|---|---|
| Figure 2: | Schematic of the saRNA Replicon for AAHI-SC2 | 23 |
| Figure 3: | Nanostructured Lipid Carrier (NLC) Schematic | 24 |
| Figure 4: | Total IgG Titers by ELISA | 26 |
| Figure 5: | AAHI-SC2 Vaccine SARS-CoV-2 Variant Neutralization | 26 |
| Figure 6: | IgG Subclass Analysis by ELISA | 27 |
| Figure 7: | CD4+ and CD8+ T Cell Responses by Intracellular Cytokine Staining with Flow Cytometry | 27 |
| Figure 8: | Study Design | 28 |
| Figure 9: | Quantification of IgG Antibody | 29 |
| Figure 10: | Quantification of IgG Antibody Subclasses | 29 |
| Figure 11: | CD4 T Cell Responses to S Protein | 30 |
| | CD8 T Cell Responses to S Protein | |
| Figure 13: | Study Schema for Nonhuman Primate Evaluation of saRNA/NLC Directly Expressing Antibodies to Zika Virus | 31 |
| Figure 14: | Detection of SEAP or Zika virus Antibodies After Intramuscular Vaccination of Nonhuman Primates | 32 |
| Figure 15: | CD8 T-Cell Responses to saRNA/NLC-Delivered Cancer Neoantigen in Nonhuman Primates | 33 |
| Figure 16: | Biodistribution of Replicating Viral RNA (rvRNA) in Solid Organs on Study Day 30, 32, and 36 | 36 |
| Figure 17: | Study Schematic for Immunogenicity and Protective Efficacy of AAHI-SC2 in Nonhuman Primates | 37 |
| Figure 18: | Schematic of the saRNA Replicon for AAHI-SC3 | 39 |
| Figure 19: | IgG Antibody Responses After AAHI-SC3 Immunization (IBRX-009; 3 Weeks Post Prime and 3 Weeks Post Boost) | 40 |
| Figure 20: | CD4+ and CD8+ T Cell Responses by Intracellular Cytokine Staining with Flow Cytometry (IBRX-009; 3 weeks post boost) | 41 |
| Figure 21: | IgG Antibody Responses After AAHI-SC3 Immunization (IBRX-012; 3 Weeks Post Prime and 2 Weeks Post Boost) | 42 |
| Figure 22: | CD4+ and CD8+ T Cell Responses by Intracellular Cytokine Staining with Flow Cytometry (IBRX-012; 2 Weeks Post Boost | 42 |

ImmunityBio, Inc.


## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|----------------------------------------|
| β-НСС | β-Human chorionic gonadotropin |
| ACE2 | Angiotensin converting enzyme 2 |
| Ad5 | Adenovirus serotype 5 |
| ARDS | Acute respiratory distress syndrome |
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| BAU | Binding antibody units |
| BSL | Biosafety level |
| BUN | Blood urea nitrogen |
| CAP | College of American Pathologists |
| CBC | Complete blood count |
| CD | Cluster of differentiation |
| CFR | Code of Federal Regulations |
| CMI | Cell mediated immunity |
| COVID-19 | Coronavirus disease 2019 |
| CRF | C se report form |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| ELISA | Enzyme linked immunosorbent assay |
| ELISpot | Enzyme linked immunosorbent spot assay |
| EOS | End of study |
| ETSD | Enhanced T cell stimulation domain |
| EUA | Emergency Use Authorization |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practices |
| GMFR | Geometric mean fold rise |
| GMT | Geometric mean titer |
| hAd5 | Human adenovirus serotype 5 |


| Abbreviation or Specialist Term | Explanation |
|---|---|
| hAd5 [E1-,E2b-,E3-] | Adenovirus serotype 5 with deletions in E1, E2b and E3 |
| hAd5-Null | Vaccine vector control with no SARS-CoV-2 antigen encoded |
| hAd5-S-Fusion+N-ETSD | Vaccine containing both full length wild type SARS-CoV-2 spike gene optimized for better spike protein expression, and full length wild type SARS-CoV-2 nucleocapsid gene modified to also contain an enhanced T cell stimulation domain (ETSD) to enhance cell-mediated immunity |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| ICF | Informed consent form |
| ICH | International Conference on Harmonization |
| ICS | Intracellular cytokine staining |
| IEC | Independent Ethics Committee |
| IFN | Interferon |
| IgG | Immunoglobulin |
| IHC | Immunohistochemistry/immunohistochemical |
| IL | Interleukin |
| IM | Intramuscular |
| IP | Investig tional product |
| IRB | Institutional Review Board |
| IUD | Intrauterine device |
| IV | Intravenous(ly) |
| LAMP | Loop-mediated isothermal amplification |
| MAAE | Medically attended adverse event |
| MoDC | Monocyte-derived dendritic cell |
| N | SARS-CoV-2 nucleocapsid antigen |
| NCI | National Cancer Institute |
| NHP | Non-human primate |
| NLC | Nanostructure lipid carrier |
| PBMC | Peripheral blood mononuclear cell |
| qPCR | Quantitative polymerase chain reaction |
| RBD | Receptor binding domain |
| RT | Reverse transcription |
| rvRNA | Replicating viral RNA |


| Abbreviation or Specialist Term | Explanation |
|---|---|
| S | SARS-CoV-2 spike antigen |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| saRNA | Self-amplifying RNA |
| SARS-CoV-2 | Severe acute respiratory syndrome coronavirus 2, the causative agent of the COVID-19 pandemic |
| SC | Subcutaneous(ly) |
| SFC | Spot forming cells |
| SoC | Standard of care |
| SOP | Standard operating procedure |
| SRC | Safety Review Committee |
| TNF | Tumor necrosis factor |
| ULN | Upper limit of normal |
| US | United States |
| VE | Vaccine Efficacy |
| VP | Viral particles |
| WBC | White blood cell |

## 1. BACKGROUND AND STUDY RATIONALE



ImmunityBio, Inc.


AAHI-SC2 and AAHI-SC3





ImmunityBio, Inc.



| AAHI-SC2 and AAHI-SC3<br>Clinical Trial Protocol: COVID-4.015 Version 4 | ImmunityBio, Inc. |
|---|---|

ImmunityBio, Inc.

AAHI-SC2 and AAHI-SC3



| AAHI-SC2 and AAHI-SC3<br>Clinical Trial Protocol: COVID-4.015 Version 4 | ImmunityBio, Inc |
|---|---|









ImmunityBio, Inc.


AAHI-SC2 and AAHI-SC3

ImmunityBio, Inc.

AAHI-SC2 and AAHI-SC3




ImmunityBio, Inc.

#### 2. STUDY OBJECTIVES

#### 2.1. Phase 1

#### 2.1.1. Primary Objective

• To determine the safety and reactogenicity of homologous and heterologous vaccination with saRNA COVID-19 vaccines.

#### 2.1.2. Secondary Objective

• To determine immunogenicity of homologous and heterologous vaccination with saRNA COVID-19 vaccines, as determined by changes in humoral and cellular response.

#### 2.2. Phase 2

## 2.2.1. Primary Objective

• To determine immunogenicity of homologous and heterologous vaccination with saRNA COVID-19 vaccines, as determined by changes in humoral and cellular response.

#### 2.2.2. Secondary Objectives

• To determine the safety and reactogenicity of homologous and heterologous vaccination with saRNA COVID-19 vaccines.